CLINICAL TRIAL: NCT02868307
Title: Response Shift and Quality of Life in Patients Suffering From Schizophrenia and Their Caregivers
Acronym: SCHIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-09; 2012-A00343-40 (Other: Ansm)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient prsenting schizophrenia (Experimental)
  Interventions: Behavioral: Answering questionnaire

INTERVENTIONS:
Behavioral: Answering questionnaire

SUMMARY:
Quality of life (QoL) measurements have become an important way to evaluate the treatments and care provided to patients with schizophrenia. Understanding determinants of QoL in schizophrenia is of importance for developing effective interventions that would improve patient functional and subjective well-being. A challenge in the interpretation of QoL measures, especially in longitudinal studies, is that QoL is self-reported by the patient and might be influenced by psychological phenomena such as adaptation to illness. An important mediator of this adaptation process is a "response shift" (RS), which involves changing internal standards, values and the conceptualization of QoL. RS can be divided into three phases 1) reconceptualization (i.e., a redefinition of QoL), 2) reprioritization (i.e., a change in the importance attributed to component domains constituting QoL) and 3) recalibration (i.e., a change in a patient's internal standards of measurements). Patients may change their frame of reference, rendering scores from different measurement occasions incomparable. An RS is a potential explanation when the QoL of an individual who has experienced a serious health event or chronic condition is similar to the QoL of a healthy individual. With an RS, the concept of QoL changes over time and cannot be compared longitudinally because of changes in internal standards, values, and/or concepts. True change may be over- or underestimated when a RS is present, leading to biased estimates of the magnitude of change.The objective is to examine whether a response shift, a change in the internal standards of a patient, occurs in patients suffering from schizophrenia and in their caregivers.

This is a monocentric and propective design study, with inclusion of patients and caregivers on a 12-month period, and a follow up on a 12-month period.

100 patients with schizophrenia and 100 caregivers

Test approach (Response shift (RS) (pre-test - then-test), unadjusted effect (post-test - pre-test), and adjusted effect (post-test - then-test scores)) will be completed with other statistical approaches such as confirmatory factorial analysis, multilevel models and CART method.

ELIGIBILITY:
Inclusion Criteria Caregiver::

* Person identified by the patient as the family member or friend who provided the most support or assistance,
* Informed consent obtained
* Being a native French speaker

Inclusion criteria patients:

* Suffering of schizophrenia according DSM IV,
* Informed consent obtained
* Being a native French speaker

Exclusion Criteria:

* Patient suffuring of demencia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of response shift occuring in patients suffering from schizophrenia and in their caregivers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Laurent BOYER, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France